CLINICAL TRIAL: NCT04559061
Title: Clinical Validation of the Vektor Computational ECG Mapping System (vMap™) for Atrial and Ventricular Arrhythmias/Pacing
Brief Title: Vektor vMap™ Clinical Validation Study
Status: Completed | Type: Observational
Sponsor: Vektor Medical (Industry)
Collaborators: Experien Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-PR-1010
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation; Ventricular Arrythmia; Premature Ventricular Complexes Multiple; Ventricular Tachycardia; Ventricular Fibrillation; Premature Atrial Complex; Atrioventricular Reentrant Tachycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Tachycardia, Ventricular; Ventricular Fibrillation; Atrial Premature Complexes; Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Cardiac ablation procedure — Retrospective data will be collected from cases where successful ablation was completed.

SUMMARY:
This is a retrospective, multi center clinical study collecting existing, de-identified subject data from medical records to be analyzed using an independent core laboratory to validate performance of a computational ECG mapping system (vMap™).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has one of the following clinical arrhythmia/pacing types:

   * Atrial pacing
   * Atrial fibrillation
   * Ventricular pacing
   * Premature ventricular complex
   * Ventricular tachycardia
   * Ventricular fibrillation
   * Focal atrial tachycardia
   * Premature atrial complex
   * Atrioventricular reentrant tachycardia
2. Patient has undergone 'successful' routine, standard of care diagnostic electrophysiology (EP) study using intracardiac catheters as clinically indicated, guided by fluoroscopy and routine electroanatomic mapping, intracardiac echocardiography, and/or cardiac imaging such as CT or MRI.
3. Patient has 12 lead electrogram data of clinical rhythms recorded on electrogram recording system.
4. Patient has undergone a successful ablation procedure.
5. Arrhythmia type and atrial/ventricular characteristics can be abstracted from patient medical records.
6. Patient was between 22 and 100 years of age at time of EP study and ablation procedure.

Exclusion Criteria:

Patients with unstable coronary artery disease, confirmed intracardiac thrombus, active sepsis, complex congenital heart disease, dextrocardia, severe pulmonary hypertension, decompensated heart failure, a mechanical heart valve, myocardial infarction within 1 month of ablation, inability to induce arrhythmia, unacceptable ECG data quality, and/or data included in the device training dataset.

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cardiac arrhythmia that have undergone successful ablation procedures.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Rate of accuracy/agreement of vMap™ in correctly identifying the ventricular chamber/region of the arrhythmia for PCV and VT. | Immediately post ablation procedure through approximately 6 months post ablation procedure, based on retrospective data collection eligibility criteria.

SECONDARY OUTCOMES:
Rate of accuracy/agreement of vMap™ in correctly identifying the chamber/region of the arrhythmia location for all arrhythmia types. | Immediately post ablation procedure through approximately 6 months post ablation procedure, based on retrospective data collection eligibility criteria.
Rate of accuracy/agreement of vMap™ in correctly identifying the segment of the arrhythmia treatment across all arrhythmia types. | Immediately post ablation procedure through approximately 6 months post ablation procedure, based on retrospective data collection eligibility criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Villongco, PhD, Study Chair — Vektor Medical
Locations (4):
- United States (4):
  - Medical University of South Carolina, Charleston, California
  - University of California San Diego Health, La Jolla, California
  - VA San Diego Healthcare System, San Diego, California
  - Sutter Health, San Francisco, California

REFERENCES:
- [Derived] Krummen DE, Villongco CT, Ho G, Schricker AA, Field ME, Sung K, Kacena KA, Martinson MS, Hoffmayer KS, Hsu JC, Raissi F, Feld GK, McCulloch AD, Han FT. Forward-Solution Noninvasive Computational Arrhythmia Mapping: The VMAP Study. Circ Arrhythm Electrophysiol. 2022 Sep;15(9):e010857. doi: 10.1161/CIRCEP.122.010857. Epub 2022 Sep 7. PMID 36069189